CLINICAL TRIAL: NCT04589676
Title: Developing and Testing the Opioid Rapid Response System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Prevention, LLC (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Principal Investigator, Michael Hecht, President, Real Prevention, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R41DA053078-01 (NIH)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Opioid Overdose
Keywords: Naloxone
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Intervention Model Description: An unblinded, two-arm, parallel group cluster-randomized trial with non-random cluster sampling will be conducted in two Indiana counties to establish the usability and feasibility of ORRS and its recruitment and training components.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal recruitment (Active Comparator): Participants in this training condition will receive recruitment messages that appeal to their personal sense of identity (e.g., you could be a hero if you get trained with naloxone).
  Interventions: Behavioral: Naloxone training
- Online training (Experimental): Participants in this training condition will receive recruitment messages that appeal to their communal sense of identity (e.g., your family and friends will thank you for getting trained with naloxone).
  Interventions: Behavioral: Naloxone training

INTERVENTIONS:
Behavioral: Naloxone training — The naloxone training will teach participants about how to appropriately use naloxone in the event of an opioid overdose.

SUMMARY:
This Phase I SBIR will develop and demonstrate the usability/feasibility of the Opioid Rapid Response System (OSSR) in order to reduce deaths and strain on emergency response systems from opioid overdoses.

DETAILED DESCRIPTION:
Opioid overdoses exact a tremendous cost in lives and expenditures due to incredible strain on emergency response systems. Naloxone has been developed to counteract overdoses. However, the nature of these events requires a rapid response, a situation that challenges emergency responders in both lightly populated rural areas as well as densely populated urban communities. PulsePoint has developed an app with the potential to obviate both concerns by linking responders to events through the 911 system. PulsePoint is already in place in 4,000 communities throughout the U.S. However, the app cannot accomplish these goals without being used by a large number of citizen responders who are both able to administer life-saving Naloxone and confident in their ability to do so. This project is designed to develop innovative and effective techniques for filling this gap. We build off of the Clark County Pilot Project conducted by members of our team that developed preliminary recruitment and training protocols for enabling citizen responders to utilize the PulsePoint App. Using communication theory, a technology-based recruitment protocol will be built around appeals to individuals (personal identity appeals) and others (communal appeals). Recruitment messages will be disseminated through diverse media channels, including social media, posters, radio announcement, and work-of-mouth. Social Cognitive Theory will be used to develop both online and face-to-face training to enable users to use the PulsePoint App, safely respond to calls, and administer Naloxone. An unblinded, two-arm, parallel group cluster-randomized trial with non-random cluster sampling will be conducted in two Indiana counties to establish the usability and feasibility of ORRS and its recruitment and training components. We anticipate recruiting and training 400 citizen responders. Pretest and posttest surveys will evaluate the training and as well as recruitment exposure through the various channels. County-level data on the number of events to which participant responded as well as lives saved also will be used to evaluate the intervention. A quasi-experimental design will compare the two recruitment strategies and the two training modalities. Project findings will be used to design and more extensive, two statewide evaluation studies (Indiana and Washington) that examine outcomes in numbers of lives saves as well as conducted a cost effectiveness analyses. The project has great promise for rapid and wide dissemination through the PulsePoint network of communities and has the potential to develop a model for community responses to similar public health events (e.g., coronavirus, stroke, heart failure).

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy citizen volunteers, aged 18 and over, living in Boone and Hancock Counties of Indiana.
* Able to understand/complete questionnaires, recruitment messages, and training procedures in English.

Exclusion Criteria:

* Those who have a Boone or Hancock County residential address, but temporarily live in another county or State, so are unable to attend training if assigned to face-to-face naloxone training.
* Those who participate in other research studies which require activities that interfere with the measurements of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Scale to measure perceptions of training program | 3 months
  Self report survey scale to measure perceptions of training using agree-disagree scale that yields a composite score of rating that the training is worth the investment of their time and they would recommend it to others in their community.

SECONDARY OUTCOMES:
Scales to measure knowledge gained from training | 3 months
  Self report on 10, multiple choice items to measure the knowledge about opioids and other information taught during training content. Scores reflect the amount of learning from training.
Scale to measure perceptions of efficacy in delivering naloxone. | 3 months
  Self report scales will measure response efficacy (i.e., administering Naloxone is effective) and self efficacy (i.e., they can administer Naloxone) using agree-disagree scales. Each subscale will consist of at least 3 items and be modified from existing efficacy scales used in drug prevention research.
Scale to measure exposure to recruitment campaign | 3 months
  Will be adapted from the evaluation of the ONCDP's substance use prevention campaigns to measure if participants recall receiving messages and the channel that they received it in. Response items will include "definitely seen", "might have seen" and "definitely not seen"

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hecht, PhD, Principal Investigator — REAL Prevention
Locations (2):
- United States (2):
  - Indiana University, Bloomington, Indiana
  - REAL Prevention LLC, Clifton, New Jersey

IPD SHARING:
Plan to Share IPD: No
Confidential data cannot be shared.

REFERENCES:
- [Background] Boslett AJ, Denham A, Hill EL. Using contributing causes of death improves prediction of opioid involvement in unclassified drug overdoses in US death records. Addiction. 2020 Jul;115(7):1308-1317. doi: 10.1111/add.14943. Epub 2020 Feb 27. PMID 32106355
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Joudrey PJ, Edelman EJ, Wang EA. Drive Times to Opioid Treatment Programs in Urban and Rural Counties in 5 US States. JAMA. 2019 Oct 1;322(13):1310-1312. doi: 10.1001/jama.2019.12562. PMID 31573628
- [Background] Cosby AG, McDoom-Echebiri MM, James W, Khandekar H, Brown W, Hanna HL. Growth and Persistence of Place-Based Mortality in the United States: The Rural Mortality Penalty. Am J Public Health. 2019 Jan;109(1):155-162. doi: 10.2105/AJPH.2018.304787. Epub 2018 Nov 29. PMID 30496008
- [Background] Compton WM, Jones CM, Baldwin GT. Relationship between Nonmedical Prescription-Opioid Use and Heroin Use. N Engl J Med. 2016 Jan 14;374(2):154-63. doi: 10.1056/NEJMra1508490. No abstract available. PMID 26760086
- [Background] Chen Q, Larochelle MR, Weaver DT, Lietz AP, Mueller PP, Mercaldo S, Wakeman SE, Freedberg KA, Raphel TJ, Knudsen AB, Pandharipande PV, Chhatwal J. Prevention of Prescription Opioid Misuse and Projected Overdose Deaths in the United States. JAMA Netw Open. 2019 Feb 1;2(2):e187621. doi: 10.1001/jamanetworkopen.2018.7621. PMID 30707224
- [Background] Flood-Grady E, Clark VC, Bauer A, Morelli L, Horne P, Krieger JL, Nelson DR. Evaluating the Efficacy of a Registry linked to a Consent to Re-Contact Program and Communication Strategies for Recruiting and Enrolling Participants into Clinical Trials. Contemp Clin Trials Commun. 2017 Dec;8:62-66. doi: 10.1016/j.conctc.2017.08.005. Epub 2017 Aug 24. PMID 29503877
- [Background] Lewis CR, Vo HT, Fishman M. Intranasal naloxone and related strategies for opioid overdose intervention by nonmedical personnel: a review. Subst Abuse Rehabil. 2017 Oct 11;8:79-95. doi: 10.2147/SAR.S101700. eCollection 2017. PMID 29066940
- [Background] Krieger JL, Palmer-Wackerly A, Dailey PM, Krok-Schoen JL, Schoenberg NE, Paskett ED. Comprehension of Randomization and Uncertainty in Cancer Clinical Trials Decision Making Among Rural, Appalachian Patients. J Cancer Educ. 2015 Dec;30(4):743-8. doi: 10.1007/s13187-015-0789-0. PMID 25608719
- [Background] Ray AE, Greene K, Hecht ML, Barriage SC, Miller-Day M, Glenn SD, Banerjee SC. An E-Learning Adaptation of an Evidence-Based Media Literacy Curriculum to Prevent Youth Substance Use in Community Groups: Development and Feasibility of REAL Media. JMIR Form Res. 2019 May 9;3(2):e12132. doi: 10.2196/12132. PMID 31094328
- [Background] Hecht ML, Marsiglia FF, Elek E, Wagstaff DA, Kulis S, Dustman P, Miller-Day M. Culturally grounded substance use prevention: an evaluation of the keepin' it R.E.A.L. curriculum. Prev Sci. 2003 Dec;4(4):233-48. doi: 10.1023/a:1026016131401. PMID 14598996
- [Background] Choi HJ, Krieger JL, Hecht ML. Reconceptualizing efficacy in substance use prevention research: refusal response efficacy and drug resistance self-efficacy in adolescent substance use. Health Commun. 2013;28(1):40-52. doi: 10.1080/10410236.2012.720245. PMID 23330857
- [Derived] Hecht ML, Jayawardene W, Henderson C, Pezalla A, Flood-Grady E, Krieger JL, Frederick A, Parker M, Ables E. Developing the Opioid Rapid Response System for Lay Citizen Response to the Opioid Overdose Crisis: a Randomized Controlled Trial. Prev Sci. 2023 Oct;24(7):1386-1397. doi: 10.1007/s11121-023-01588-0. Epub 2023 Sep 22. PMID 37737966
- [Derived] Jayawardene W, Pezalla A, Henderson C, Hecht M. Development of opioid rapid response system: Protocol for a randomized controlled trial. Contemp Clin Trials. 2022 Apr;115:106727. doi: 10.1016/j.cct.2022.106727. Epub 2022 Mar 13. PMID 35296414
- See also: Related Info — https://www.cdc.gov/drugoverdose/index.html